CLINICAL TRIAL: NCT05121688
Title: Effectiveness of a Multimodal Physical Therapy Telerehabilitation Program in Long Post COVID-19 Symptoms in Primary Health Care.
Brief Title: Effectiveness of a Physical Therapy Telerehabilitation Program in Long Post COVID-19 Symptoms in Primary Health Care.
Acronym: TPhysioCovid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Spanish Primary Health Care (Unknown)
Responsible Party: Principal Investigator, MARIA JOSE DIAZ ARRIBAS, University Professor, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCMadrid
Record Dates: First submitted 2021-11-10; First posted 2021-11-16 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: COVID-19; Physical Therapy Modalities; Telerehabilitation; Primary Health Care
Keywords: COVID-19; Physical Therapy; Telerehabilitation; Primary Health Care
MeSH Terms: conditions — COVID-19 | interventions — Physical Therapy Modalities; Exercise Therapy

STUDY DESIGN:
Intervention Model Description: The participants will be randomly allocated to Tele-physiotherapy or control groups.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The Principal Investigator and the assessor will be blinded to the randomization and allocation. The assessor will have not access to patients' medical record. Patients will be also asked to do not explain about their procedure to the assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-physiotherapy group (Experimental): Allocated participants to intervention group will receive 18 Tele-physiotherapy sessions (three sessions per week, with 30 min. of duration) during six weeks. In this sessions, participants will carry out a tele-face-to-face multimodal physical therapy program based on health education, respiratory exercises, physical training exercises, aerobic exercises and functional mobility.
  This group will receive conventional medical care too.
  Interventions: Other: Physiotherapy
- Control group (Active Comparator): No Physical therapy intervention. Allocated participants to control group will receive one consultation session by the physiotherapist, but will not received any physical Therapy treatment. At this session, patients will be educated about how to perform their daily activities, breathing exercises, walking. Conventional medical care will be provided.
  In the control group, the same measurements will be made at the same times as the subjects in the intervention group. Once the study is finished, the researcher agrees to carry out the intervention to the patients in the control group.
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy — A Tele-face-to-face multimodal physical therapy program based on health education, respiratory exercises, physical training exercises, aerobic exercises and functional mobility.
  Other Names: Therapeutic exercise

SUMMARY:
The evolution of Coronavirus disease 2019 (COVID-19) pandemic makes it more necessary the intervention of Primary Health Care Physiotherapy Units in patients with respiratory and/or functional sequelae after suffering from SARS-CoV-2 (acute respiratory sindrome by coronavirus) virus infection.

Since some months ago, Primary Health Care use telerehabilitation tools to connect patients and health care professions while maintaining social distancing and restrictions. Tele-physiotherapy is a field of physiotherapy which has the advantage of providing physical therapy interventions to patients' complications after COVID-19 by using a videoconferencing method. The aim of this study is to evaluate the effectiveness of a multimodal Physical Therapy telerehabilitation program in persistent post COVID-19 symptoms in Primary Health Care.

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19), is a multisystem infectious disease which has led to a global pandemic. The evolution of COVID-19 disease makes it more necessary the intervention of Primary Health Care Physiotherapy Units in patients with respiratory and /or functional sequelae after suffering from SARS-CoV-2 infection. Problems such as breathlessness, exercise intolerance and loss of peripheral muscle strength can be observed in individuals who have been diagnosed with persistent post COVID-19.

Since some months ago, Primary Health Care use telerehabilitation tools to connect patients and health care professions while maintaining social distancing and restrictions. Tele-physiotherapy is a field of physiotherapy which has the advantage of providing physical therapy interventions to patients' complications after COVID-19 by using a videoconferencing method. The aim of this study is to evaluate the effectiveness of a multimodal Physical Therapy telerehabilitation program in persistent post COVID-19 symptoms in Primary Health Care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with long post-COVID symptoms (from week 12 to week 24).
* Patients between 25 and 70 years old.
* Patients with moderate respiratory and/or functional affectation with long post COVID-19 symptoms, belonging to four Physiotherapy Units of primary Health Care in Madrid (Spain).
* Confirmed diagnosis of COVID-19 via a positive nasopharyngeal or throat swab within the past 12 months.
* Persistent symptoms lasting ≥12 weeks since the first positive test, including dyspnea (new or increased from baseline as measured by modified Medical Research Council (mMRC) score ≥1).
* Normal oxygen saturation (greater than 90%) by pulse oximetry at rest on room air.
* Participant owns a smart phone, tablet, or computer to access on-line sessions.

Exclusion Criteria:

* People with symptoms such as fever, cough, upper respiratory distress, diarrhea, vomiting, anosmia or ageusia.
* Temperature greater than 37.2 degrees Celsius.
* Patients with multimorbidity. Multimorbidity will be considered when the patient is diagnosed with two or more diseases among the following: diabetes, dyslipidaemia, cardiovascular disease (arterial hypertension, ischemic heart disease, valvular heart disease, heart failure), osteoarthritis, respiratory disease (asthma, chronic bronchitis), digestive disease ( gastric or duodenal ulcers, inflammatory bowel disease, liver disease), psychiatric pathology or tumor pathology.
* Patients with previous pathologies: ischemic heart disease, dementia, lung failure, lung cancer, cystic fibrosis, pulmonary fibrosis, chronic kidney failure, liver diseases, myocardial arrhythmias, deep vein thrombosis, severe aortic stenosis, liver diseases.
* Patients with weakened immune systems: in cancer treatment, organ or marrow transplant patients, HIV/AIDS, prolonged use of prednisone or similar medication.
* Patients with functional limitations to carry out their basic activities of daily living. Barthel index greater than 90.
* Patients with cognitive problems. Mini-Cognitive Lobo exam greater than 23 points
* Active bleeding.
* Unstable fractures.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2021-11-25 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2023-05-09 (Actual)

PRIMARY OUTCOMES:
Modified Borg scale. | Baseline.
  Modified Borg scale, or scale of perceived exertion, is a subjective scale to measure the intensity of a physical effort, quantifying the respiratory distress. The modified Borg Scale is averaged from 0 to 10. Perceived effort will be measured as 0-2 (light effort), 3-4 (moderate effort), 5-6 (hard effort), 7-9 (very hard effort) and 10 (maximum effort).
Modified Borg scale. | 6 weeks.
  Modified Borg scale, or scale of perceived exertion, is a subjective scale to measure the intensity of a physical effort, quantifying the respiratory distress. The modified Borg Scale is averaged from 0 to 10. Perceived effort will be measured as 0-2 (light effort), 3-4 (moderate effort), 5-6 (hard effort), 7-9 (very hard effort) and 10 (maximum effort).
Modified Borg scale. | 10 weeks.
  Modified Borg scale, or scale of perceived exertion, is a subjective scale to measure the intensity of a physical effort, quantifying the respiratory distress. The modified Borg Scale is averaged from 0 to 10. Perceived effort will be measured as 0-2 (light effort), 3-4 (moderate effort), 5-6 (hard effort), 7-9 (very hard effort) and 10 (maximum effort).
Modified Borg scale. | 14 weeks.
  Modified Borg scale, or scale of perceived exertion, is a subjective scale to measure the intensity of a physical effort, quantifying the respiratory distress. The modified Borg Scale is averaged from 0 to 10. Perceived effort will be measured as 0-2 (light effort), 3-4 (moderate effort), 5-6 (hard effort), 7-9 (very hard effort) and 10 (maximum effort).

SECONDARY OUTCOMES:
Modified Medical Research Council Dyspnea Score. | Baseline.
  Modified Medical Research Council Dyspnea Score (mMRC). The mMRC Dyspnea Score is used to establish baseline functional impairment due to dyspnea.The severity of dyspnea is rated on a scale of 0 to 4. "O" means no dyspnea perception, "4" means severe dyspnea perception.
  Grade 0: absence of dyspnea when performing intense exercise. Grade 1: dyspnea when walking quickly on the flat or climbing. Grade 2: dyspnea does not allow walking with another person of the same age or the person has to stop to rest.
  Grade 3: dyspnea makes the patient stops to rest when walking for 100m or a few minutes after walking on the flat.
  Grade 4: dyspnea prevents the patient from leaving home or appears in activities of daily living.
Modified Medical Research Council Dyspnea Score. | 6 weeks.
  Modified Medical Research Council Dyspnea Score (mMRC). The mMRC Dyspnea Score is used to establish baseline functional impairment due to dyspnea.The severity of dyspnea is rated on a scale of 0 to 4. "O" means no dyspnea perception, "4" means severe dyspnea perception.
  Grade 0: absence of dyspnea when performing intense exercise. Grade 1: dyspnea when walking quickly on the flat or climbing. Grade 2: dyspnea does not allow walking with another person of the same age or the person has to stop to rest.
  Grade 3: dyspnea makes the patient stops to rest when walking for 100m or a few minutes after walking on the flat.
  Grade 4: dyspnea prevents the patient from leaving home or appears in activities of daily living.
Modified Medical Research Council Dyspnea Score. | 10 weeks.
  Modified Medical Research Council Dyspnea Score (mMRC). The mMRC Dyspnea Score is used to establish baseline functional impairment due to dyspnea.The severity of dyspnea is rated on a scale of 0 to 4. "O" means no dyspnea perception, "4" means severe dyspnea perception.
  Grade 0: absence of dyspnea when performing intense exercise. Grade 1: dyspnea when walking quickly on the flat or climbing. Grade 2: dyspnea does not allow walking with another person of the same age or the person has to stop to rest.
  Grade 3: dyspnea makes the patient stops to rest when walking for 100m or a few minutes after walking on the flat.
  Grade 4: dyspnea prevents the patient from leaving home or appears in activities of daily living.
Modified Medical Research Council Dyspnea Score. | 14 weeks.
  Modified Medical Research Council Dyspnea Score (mMRC). The mMRC Dyspnea Score is used to establish baseline functional impairment due to dyspnea.The severity of dyspnea is rated on a scale of 0 to 4. "O" means no dyspnea perception, "4" means severe dyspnea perception.
  Grade 0: absence of dyspnea when performing intense exercise. Grade 1: dyspnea when walking quickly on the flat or climbing. Grade 2: dyspnea does not allow walking with another person of the same age or the person has to stop to rest.
  Grade 3: dyspnea makes the patient stops to rest when walking for 100m or a few minutes after walking on the flat.
  Grade 4: dyspnea prevents the patient from leaving home or appears in activities of daily living.
Saint George Respiratory Questionnaire. | Baseline.
  Saint George Respiratory Questionnaire (SGRQ) is a questionnaire to assess the quality of life in patients with respiratory problems. It is made up of 50 items divided into three scales: symptoms, activity and impact. The SGRQ ranges from 0 (no impairment of quality of life) to 100 (highest impairment of quality of life).
Saint George Respiratory Questionnaire. | 6 weeks.
  Saint George Respiratory Questionnaire (SGRQ) is a questionnaire to assess the quality of life in patients with respiratory problems. It is made up of 50 items divided into three scales: symptoms, activity and impact. The SGRQ ranges from 0 (no impairment of quality of life) to 100 (highest impairment of quality of life).
Saint George Respiratory Questionnaire. | 10 weeks.
  Saint George Respiratory Questionnaire (SGRQ) is a questionnaire to assess the quality of life in patients with respiratory problems. It is made up of 50 items divided into three scales: symptoms, activity and impact. The SGRQ ranges from 0 (no impairment of quality of life) to 100 (highest impairment of quality of life).
Saint George Respiratory Questionnaire. | 14 weeks.
  Saint George Respiratory Questionnaire (SGRQ) is a questionnaire to assess the quality of life in patients with respiratory problems. It is made up of 50 items divided into three scales: symptoms, activity and impact. The SGRQ ranges from 0 (no impairment of quality of life) to 100 (highest impairment of quality of life).
6-Minute Walk Test (6MWT). | Baseline.
  6MWT is a test that measures the distance walked by each patient for 6 minutes, 30 meters on a flat and hard surface. The 6MWT assesses the level of submaximal functional capacity. The patient has to walk as far as possible for 6 minutes.
  Performance is classified into 4 categories:
  Category A: less than 350 meters; poor performance. Category B: between 350 and 450 meters; moderate performance. Category C: between 450 and 650 meters; good performance. Category D: more than 650 meters; excellent performance.
6-Minute Walk Test (6MWT). | 6 weeks.
  6MWT is a test that measures the distance walked by each patient for 6 minutes, 30 meters on a flat and hard surface. The 6MWT assesses the level of submaximal functional capacity. The patient has to walk as far as possible for 6 minutes.
  Performance is classified into 4 categories:
  Category A: less than 350 meters; poor performance. Category B: between 350 and 450 meters; moderate performance. Category C: between 450 and 650 meters; good performance. Category D: more than 650 meters; excellent performance.
6-Minute Walk Test (6MWT). | 10 weeks.
  6MWT is a test that measures the distance walked by each patient for 6 minutes, 30 meters on a flat and hard surface. The 6MWT assesses the level of submaximal functional capacity. The patient has to walk as far as possible for 6 minutes.
  Performance is classified into 4 categories:
  Category A: less than 350 meters; poor performance. Category B: between 350 and 450 meters; moderate performance. Category C: between 450 and 650 meters; good performance. Category D: more than 650 meters; excellent performance.
6-Minute Walk Test (6MWT). | 14 weeks.
  6MWT is a test that measures the distance walked by each patient for 6 minutes, 30 meters on a flat and hard surface. The 6MWT assesses the level of submaximal functional capacity. The patient has to walk as far as possible for 6 minutes.
  Performance is classified into 4 categories:
  Category A: less than 350 meters; poor performance. Category B: between 350 and 450 meters; moderate performance. Category C: between 450 and 650 meters; good performance. Category D: more than 650 meters; excellent performance.

CONTACTS AND LOCATIONS:
Overall Officials: María José Díaz-Arribas, PhD., Principal Investigator — Director of Physical Therapy Section.; Gustavo Plaza Manzano, PhD., Study Director — Sub-director of Pysical Therapy Section.; Mabel Ramos Sánchez, PhD., Study Director — Tenured University Professor.; José Calvo Paniagua, Master, Principal Investigator — Associated Clinical Professor
Locations (1):
- María José Díaz Arribas, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Calvo-Paniagua J, Diaz-Arribas MJ, Valera-Calero JA, Ramos-Sanchez M, Fernandez-de-Las-Penas C, Navarro-Santana MJ, Del Corral T, Plaza-Manzano G. Educational, Exercise, and Occupational Therapy-Based Telerehabilitation Program Versus "Wait-and-See" for Improving Self-perceived Exertion in Patients With Post-COVID Fatigue and Dyspnea: A Randomized Clinical Trial. Am J Phys Med Rehabil. 2024 Sep 1;103(9):797-804. doi: 10.1097/PHM.0000000000002441. Epub 2024 Jan 31. PMID 38320238